CLINICAL TRIAL: NCT01920789
Title: A Multicenter Randomized Phase II Study of Stereotactic Hypofractionated Radiotherapy With Body Frame Versus Conventionally Fractionated Radiotherapy for Stage I Medically Inoperable Non-small Cell Lung Cancer
Brief Title: Stereotactic Precision And Conventional Radiotherapy Evaluation
Acronym: SPACE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ass. Prof. Jan Nyman (Network)
Collaborators: Göteborg University (Other); Karolinska Institutet (Other)
Responsible Party: Sponsor-Investigator, Ass. Prof. Jan Nyman, Ass. Prof. Jan Nyman, Swedish Lung Cancer Study Group
Organization: Swedish Lung Cancer Study Group (Network)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPACE
Record Dates: First submitted 2013-08-05; First posted 2013-08-12 (Estimated); Last update posted 2014-12-09 (Estimated); Status verified 2014-12

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Non-small call lung cancer; Medically inoperable; Stage one; Radiotherapy; SBRT; Hypofractionation; Conventional fractionation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stereotactic radiotherapy (Experimental): Arm A: Stereotactic radiotherapy to a dose of 66 Gy at the isocenter with 22 Gy per fraction in 3 fractions during one week with body frame fixation and a planning target volume with a 5 mm margin around the macroscopic tumour. A heterogeneous dose distribution is used so 45 Gy will cover the PTV.
  Interventions: Radiation: Stereotactic radiotherapy
- Conventionally fractionated radiotherapy (Active Comparator): Arm B: Conventionally fractionated radiotherapy to a dose of 70 Gy with 2 Gy per fraction in 35 fractions during 7 weeks with fixation in a vacuum pillow and a planning target volume with a 2 cm margin around the macroscopic tumour.
  Interventions: Radiation: Conventionally fractionated radiotherapy

INTERVENTIONS:
Radiation: Stereotactic radiotherapy — Margin between CTV and PTV of 5 mm in transversal direction (except for small targets (<3cm) not fixed to thoracic wall or mediastinal structures, where margin should be 10 mm) and 10 mm in longitudinal direction. Planned heterogeneous dose distribution within the PTV with about 50% higher dose to the center compared to the periphery. Hypofractionation with 22 Gy times 3 at the isocenter (15 Gy at the periphery of the PTV)during one week will be used.
  Arms: Stereotactic radiotherapy
Radiation: Conventionally fractionated radiotherapy — Clinical target volume (CTV) comprises the Gross Tumor Volume (GTV), including its diffuse growth at the borders. Planning target volume (PTV) is defined as the CTV with a total margin of 2 cm in all directions. The patient will receive 35 fractions, with a dose of 2.0 Gy/fraction at the ICRU reference point to a total dose of 70 Gy. The treatments will be given five days a week. The total treatment time should be as close to seven weeks as possible. The aim is that the dose distribution should be as homogeneous as possible.
  Arms: Conventionally fractionated radiotherapy

SUMMARY:
A randomized phase II study for medically inoperable stage I non-small cell lung cancer where stereotactic body radiotherapy in three fractions to 66 Gy is compared with conventionally fractionated radiotherapy to 70 Gy in 35 fractions.

DETAILED DESCRIPTION:
This is a multicenter Scandinavian randomized phase II study of stereotactic hypofractionated radiotherapy with body frame versus conventionally fractionated radiotherapy for stage I medically inoperable non-small cell lung cancer patients. There is a 1:1 randomization between arm A: Stereotactic radiotherapy to a dose of 66 Gy with 22 Gy per fraction at the isocenter (45 Gy covers the PTV) in 3 fractions during one week with body frame fixation and a planning target volume with a 5 mm margin around the macroscopic tumour, and arm B: Conventionally fractionated radiotherapy to a dose of 70 Gy with 2 Gy per fraction in 35 fractions during 7 weeks with fixation in a vacuum pillow and a planning target volume with a 2 cm margin around the macroscopic tumour.

ELIGIBILITY:
Inclusion Criteria:

* Non-small cell lung cancer stage I: T1-2 N0 M0.
* Medically inoperable patients or patients refusing surgery.
* Morphologically verified. If that is impossible there must be increased tumour size in repeated CT scans and positive PET.
* Patients should have a life expectancy of > 6 months.
* WHO performance status 0-2.
* Signed written informed consent obtained.
* Patient should be feasible for both study arms.

Exclusion Criteria:

* Patients with central tumour growth adjacent to trachea, main bronchus or esophagus.
* Maximal tumour diameter > 6 cm.
* Patients with prior malignancy within the last five years (except basal cell carcinoma of the skin or in situ carcinoma of the cervix).
* Any prior antitumoral treatment of the present lung cancer.
* Previous irradiation that included part of the lung.
* Pregnant women.

Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2007-01; Primary Completion 2015-03 (Estimated); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
Freedom from tumor progression | At 36 months after randomization
  complete remission,partial remission or stable disease

SECONDARY OUTCOMES:
Overall survival | At 36 monts after randomization

OTHER OUTCOMES:
Toxicity | At 7 weeks, 3, 6, 12, 18, 24 and 36 months after randomization
  CTC version 3.0 will be used for acute and late toxicity
Quality of life | At 7 weeks, 6 and 24 months after randomization
  EORTC QLQ 30 + LC 14 questionnaire will be used

CONTACTS AND LOCATIONS:
Overall Officials: Jan Nyman, Ass. Prof, Principal Investigator — Department of Oncology, Sahlgrenska University Hospital